CLINICAL TRIAL: NCT00003095
Title: S9719: Clonal Hematopoiesis as a Marker of Genetic Damage Following Adjuvant Chemotherapy for Breast Cancer: Pilot Study to Evaluate Incidence. Ancillary to S9623
Brief Title: S9719 Gene Damage Following Chemotherapy in Women With Stage II or Stage III Breast Cancer
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000065813; S9719 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-05-19 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage III breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- bone marrow transplant: bone marrow transplant
- standard chemotherapy: standard chemotherapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy for breast cancer may damage the genes of cells. This may lead to the development of secondary cancers.

PURPOSE: Pilot study to evaluate the degree of gene damage following chemotherapy in women with stage II or stage III breast cancer involving four to nine axillary lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the incidence of early genetic damage, defined by the presence of clonal hematopoiesis using the human androgen receptor assay (HUMARA), in pretreatment blood and bone marrow, apheresis, and two sequential post-treatment specimens from women with stage II/III breast cancer enrolled in SWOG-S9623. II. Detect genetic damage following dose-intensive adjuvant regimens for breast cancer by screening for the presence of defective DNA mismatch repair mechanisms and loss of heterozygosity using microsatellite instability assays. III. Estimate the incidence of myeloid lymphoid leukemia gene fusion transcripts in cases where either the HUMARA or microsatellite repeat assays are positive for clonal hematopoiesis. IV. Determine the frequency of RAS gene mutations (H-, K-, and N-RAS) following dose-intensive adjuvant regimens for breast cancer.

OUTLINE: Prior to beginning treatment on SWOG-9623, blood samples and bone marrow aspirates (when available) are collected from each patient. Patients randomized to autologous peripheral stem cell transplant have specimens collected again at 3 months (apheresis aliquot and blood). At 3 and 12 months after completing chemotherapy, blood samples are collected from all patients. Samples are collected again from any patient presenting with a second malignancy in the future. DNA is collected from blood or bone marrow samples. Clonality at the HUMARA locus is examined. Microsatellite instability is assessed at multiple chromosomal loci: 7q31, 5q31, 17p12, 8p22, 11q23, and the BAT loci. If the HUMARA or microsatellite repeat assays are positive for clonal hematopoiesis, then specimens are examined for myeloid lymphoid leukemia fusion transcripts commonly reported in acute myeloid leukemia with 11q23 abnormalities. Specimens are also examined for RAS mutations (H-, K-, N-RAS). Patients do not receive the results of the genetic testing and the results do not influence the type or duration of treatment.

PROJECTED ACCRUAL: This study will accrue 100 patients for each arm of SWOG-9623, for a total of 200 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Must be enrolled in SWOG-9623 at time of registration to this study, but must not have started treatment Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Adult Sex: Female Menopausal status: Not specified Performance status: See Disease Characteristics Life expectancy: SWOG 0 or 1 Hematopoietic: See Disease Characteristics Hepatic: See Disease Characteristics Renal: See Disease Characteristics

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Must be enrolled in SWOG-9623 at time of registration to this study, but must not have started treatment Hormone receptor status: Not specified
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 1997-11; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn L. Slovak, PhD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (83):
- United States (83):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington